CLINICAL TRIAL: NCT04507945
Title: The Goal-direct Treatment of Chronic Bowel Dysfunction
Brief Title: Stablishment of Prevention and Treatment System for Intestinal Dysfunction
Acronym: A
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Lei Zheng, General surgery, Nanjing University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Intestinal dysfunction
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Intestinal dysfunction is defined as the damage of intestinal substance and/or function, which leads to digestion, absorption and/or mucosal barrier function.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- living quality (Experimental)
  Interventions: Drug: Nutritional Therapy, Metabolic Disorder, Regular
- complication (Experimental)
  Interventions: Drug: Nutritional Therapy, Metabolic Disorder, Regular

INTERVENTIONS:
Drug: Nutritional Therapy, Metabolic Disorder, Regular — According to the result reported by Byrne, Wilmore, etc. in 1992 ~ 1995, the use of growth hormone, glutamine, modified diet and other measures proposed intestinal rehabilitation treatment. Then, check the patient's quality of life survey, nutritional status, inflammation indicators and other changes every three months, and use metabolomics and microbiomic tools to detect changes in the patient's nutritional metabolism, intestinal microecology, etc., and adjust the patient's nutritional treatment and microecological treatment based on the results Program.

SUMMARY:
Dysfunction and intestinal endocrine dysfunction. This project will use genomics, metabonomics, microbiome and other omics techniques to study the clinical pathway of CID integrated therapy.

ELIGIBILITY:
Inclusion Criteria:

* The Patients with chronic bowel dysfunction

Exclusion Criteria:

* Past severe underlying diseases of the respiratory system and cardiovascular system,
* Allergy to treatment-related drugs,
* Pregnancy,
* Accept CID surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
nutrition index | 3 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pironi L, Corcos O, Forbes A, Holst M, Joly F, Jonkers C, Klek S, Lal S, Blaser AR, Rollins KE, Sasdelli AS, Shaffer J, Van Gossum A, Wanten G, Zanfi C, Lobo DN; ESPEN Acute and Chronic Intestinal Failure Special Interest Groups. Intestinal failure in adults: Recommendations from the ESPEN expert groups. Clin Nutr. 2018 Dec;37(6 Pt A):1798-1809. doi: 10.1016/j.clnu.2018.07.036. Epub 2018 Aug 18. PMID 30172658
- [Result] He D, Wang S, Hu H, Yin HY. [Advances in the research of protective effect of curcumin on intestinal mucosal barrier function]. Zhonghua Shao Shang Za Zhi. 2019 Feb 20;35(2):157-160. doi: 10.3760/cma.j.issn.1009-2587.2019.02.013. Chinese. PMID 30798584